CLINICAL TRIAL: NCT02318680
Title: Follow Home Visits by Hospital and Municipality After Discharge of Frail Elderly Patients From Nykøbing Falster Hospital - a Randomized Controlled Trial
Brief Title: Follow Home Visits After Discharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Region Zealand (Other); Nykøbing Falster County Hospital (Other); Guldborgsund Municipality (Unknown); Lolland Municipality (Unknown); Vordingborg Municipality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SJ-329
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Discharge Planning; Readmission; Hospital; Frail Elderly Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Review of follow home visits after discharge from Nykøbing Falster Hospital
  Interventions: Other: Review of follow home visits after discharge from Nykøbing Falster Hospital
- Control (No Intervention): Standard health care and discharge services

INTERVENTIONS:
Other: Review of follow home visits after discharge from Nykøbing Falster Hospital — The intervention is follow home visits which is randomized and is an intervention that is assigned by the investigator.
  Arms: Intervention

SUMMARY:
The study aims to assess whether a follow home visit after discharge of frail elderly patients from Nykøbing Falster Hospital reduces the risk of readmission within 180 days.

Staff from the hospital ward identifies patients fulfilling the inclusion criteria and refers the patients to two project nurses at the hospital (follow home team). One of the project nurses gets the informed consent from the patient, or in case of a patient who is not able to give informed consent, from the family and general practitioner. The patient is then randomized to intervention (follow home visit after discharge) or control.

In the intervention group, the hospital project nurse and the patient meets with the municipal nurse in the patient's home on the same day the patient is being discharged from the hospital. During this visit the discharge from the hospital and the actual functioning of the patient in his own surroundings is reviewed, using a structured assessment.

DETAILED DESCRIPTION:
The study consists of two parts: First, the project nurse reviews the patients hospitalization and discharge together with the nurse from the ward. Next, the patient is discharged from the hospital and is driven by the project nurse from the hospital to the patient's home where they meet the nurse from the municipality. Together with the patient the two nurses review:

* Cognitive skills
* Medicine
* Nutrition
* Mobility
* Level of functioning
* Future appointments in the health care sector

All patients in the project - both patients in the intervention group and patients in the control group - will receive treatment and care equivalent to normal applicable quality standards with discharge from the hospital.

It is expected that the study will demonstrate a reduction of hospital readmissions within 180 days in the intervention group with 14 % (with a power of 90% and a significance level of 5%). There will be a need for 200 patients in both the control and intervention group, ie 400 patients in total.

ELIGIBILITY:
Inclusion Criteria:

* Discharge from the Medical Department, Geriatric Department B, Emergency Department, Surgical Department or Department of Orthopedic Surgery at Nykøbing Falster Hospital.

Address in Guldborgsund, Lolland or Vordingborg municipalities.

Minimum 3 out of the following 9 criteria must be met:

* The patient's behavior raises suspicion of cognitive disorders, including dementia, which affects how the patient masters his daily life.
* The patient has an abuse of medication, drugs and / or alcohol, which affects how the patient masters his daily life.
* The patient has a psychiatric disorder that affects how the patient masters his daily life.
* The patient has a strained - or no - social network.
* The patient has a significantly lower level of functioning compared to prior to admission.
* The patient uses 6 or more different types of drugs at the time of discharge.
* The patient has, within the preceding 6 months, had at least one acute hospital contact beyond the current.
* The patient has a fall-history where the cause is not yet determined.
* There are suspicion of housing conditions that hamper the patient in his daily activities.

Exclusion Criteria:

* Patients who do not want to participate or cannot give informed consent. Discharge between 4 pm and 8 am Monday-Friday and discharge on weekends. Patients with planned readmission. Former participant in the study. Patients who needs terminal care.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 545 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who are readmitted | 180 days

SECONDARY OUTCOMES:
Total use of municipal services (nursing, practical help, personal care) | 180 days
The number of contacts with general practitioner | 180 days
Time to readmission | 180 days
Total number of readmissions | 180 days
Total number of days of readmission | 180 days
Death | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Antoine Lembeck, MD, Study Director — Region Zealand, Nykøbing Falster Hospital
Locations (1):
- Region Zealand, Nykøbing Falster Hospital, Nykøbing Falster, Denmark

REFERENCES:
- [Derived] Lembeck MA, Thygesen LC, Sorensen BD, Rasmussen LL, Holm EA. Effect of single follow-up home visit on readmission in a group of frail elderly patients - a Danish randomized clinical trial. BMC Health Serv Res. 2019 Oct 25;19(1):751. doi: 10.1186/s12913-019-4528-9. PMID 31653219